CLINICAL TRIAL: NCT04990141
Title: Prospective Clinical Study for the Early Detection of Preeclampsia Based on the Molecular Screening At the First Trimester of Pregnancy
Brief Title: Molecular Screening Method for Preeclampsia (PREMOM)
Acronym: PREMOM
Status: Completed | Type: Observational
Sponsor: iPremom (Industry)
Responsible Party: Sponsor
Other Study IDs: IGX1-PRE-CS-20-11
Record Dates: First submitted 2021-07-23; First posted 2021-08-04 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; Early onset Preeclampsia (EOPE); Late onset Peeclampsia (LOPE); First trimester; Early screening; Circulating RNA (C-RNA); Molecular profile; Blood
MeSH Terms: conditions — Pre-Eclampsia | interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal peripheral blood samples with circulating genetic material (C-RNA/C-DNA) and other biomolecules and cellular component to provide preeclampsia information and other obstetric complications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases group: Women recruited between 9 and 14 gestational weeks diagnosed with preeclampsia or other complication at the end of pregnancy
  Interventions: Procedure: Peripheral blood collection in cases group
- Control group: Women recruited between 9 and 14 gestational weeks without diagnosis of preeclampsia or other complication at the end of the pregnancy
  Interventions: Procedure: Peripheral blood collection in control group

INTERVENTIONS:
Procedure: Peripheral blood collection in cases group — Maternal peripheral blood will be collected 3 times during pregnancy (1st, 2nd and 3rd trimester) and clinical data compiled in cases group
  Groups: Cases group
Procedure: Peripheral blood collection in control group — Maternal peripheral blood will be collected 3 times during pregnancy (1st, 2nd and 3rd trimester) and clinical data compiled in control group
  Groups: Control group

SUMMARY:
Preeclampsia (PE) is a major obstetric complication with short- and long-term consequences for the mother and the fetus. Early screening tools to reduce its mortality and morbidity, as well as to prevent the life-threatening consequences are needed. Thus, the detection of women at risk of suffering PE is key to apply preventive and treatment strategies. Recently, the maternal contribution to PE based on defective decidualization has been evidenced and new technical approaches developed to detect circulating biomolecules in blood such as RNA fragments. The main objective of this study is to evaluate the diagnostic precision of the molecular profile from the maternal blood analysed for the early screening of early onset preeclampsia (EOPE).

DETAILED DESCRIPTION:
The hypothesis is that there is a unique molecular profile in peripheral blood specific to women who develop EOPE that allow an early assess woman´s risk of developing this pregnancy complication.

The purposed study is a biomedical, prospective, multicentre, case-control aimed to determine the predictive value and diagnostic precision of the maternal blood molecular profile for the early screening of EOPE. Late-onset preeclampsia (LOPE) and other pregnancy complications (such as preterm birth, intrauterine growth restriction, gestational diabetes, placenta previa, placental abruption, placenta accreta, premature rupture of preterm membranes, antepartum fetal death, uterine rupture and previous vasa, among others) could be analysed as a secondary outcome.

Subjects will be 9585 pregnant women recruited between 9 and 14 gestational weeks. Participants will provide peripheral blood sample at three different times during pregnancy to be characterised at molecular level in the iPremom laboratories (Igenomix Preeclampsia SLU) after their obstetric outcome was known.

Once the 50% of the total enrolment is achieved, an interim analysis will be conducted by an independent external committee. Data will be registered in an electronic Case Report Form (eCRF) specifically designed for this study. Monitoring activities and data verification will be performed during the whole study to ensure data quality, integrity and transparency.

The total estimated duration of the study is 30 months, of which the first 18 months will correspond to the recruitment period of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose written informed consent approved by the Ethics Committee (EC) has been obtained, after having been duly informed of the nature of the study and voluntarily accepted to participate after being fully aware of the potential risks, benefits and any discomfort involved.
* Women over the age of 18 at the time of signing the informed consent form.
* Pregnant women with single gestation between weeks 9 and 14 of gestation.

Exclusion Criteria:

* Known malignancy
* History of organ transplant or bone marrow transplant.
* Maternal transfusion in the last 8 weeks prior to taking the sample.
* Early gestational loss
* Existence of serious or uncontrolled bacterial, fungal or viral infections that, in the opinion of the investigator may interfere with the patient's participation in the study or the evaluation of the results of the study.
* Other circumstances or difficulties that, in the investigator's opinion, may suppose a risk to the subject or reduce the chances of obtaining satisfactory data to achieve the objectives of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women over 18 years old
Study Population: Pregnant women over the age of 18 recruited between 9 and 14 gestational weeks who attend the participating referral centers for their regular gynecological-obstetric follow-up, as well as their childbirth care.
Sampling Method: Non-Probability Sample
Enrollment: 9586 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Diagnostic precision of EOPE at molecular level | 33 weeks
  Sensitivity, specificity, positive and negative predictive value using the clinical outcome of pregnancy as a "gold standard" parameter

SECONDARY OUTCOMES:
Diagnostic precision of LOPE and other pregnancy complications at molecular level | 33 weeks
  Sensitivity, specificity, positive and negative predictive value using the clinical outcome of pregnancy as a "gold standard" parameter
Characterization of molecular profile in maternal blood | 33 weeks
  Molecular profile (DNA/RNA/proteins/metabolites) associated to gestational age, epidemiological and clinical variables

OTHER OUTCOMES:
Identification of candidate biomarkers in the maternal blood for therapy studies. | 33 weeks
  DNA/RNA/proteins/metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Garrido, PhD, Principal Investigator — iPremom (Igenomix Preeclampsia SLU)
Locations (15):
- Spain (15):
  - Hospital Universitario de Torrejón, Torrejón de Ardoz, Madrid
  - Hospital General Universitario Santa Lucía, Cartagena, Murcia
  - Hospital Universitario y Politécnico La Fe, Valencia, Valencia
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Complejo Hospitalario Universitario Insular Materno Infantil, Albacete
  - Hospital General de Alicante, Alicante
  - Hospital General de Castellón, Castellon
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital del Río Hortega, Valladolid
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No